CLINICAL TRIAL: NCT04625803
Title: Camrelizumab and Apatinib Combined With Chemotherapy (mFOLFOX6) in Neoadjuvant Therapy for Locally Advanced Colon Cancer
Brief Title: Neoadjuvant Therapy for Locally Advanced Colon Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weijia Fang, MD, Director of Medical Oncology, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMBITION
Record Dates: First submitted 2020-11-04; First posted 2020-11-12 (Actual); Results first posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: Colon Cancer; Neoadjuvant Therapy
Keywords: colon cancer; camrelizumab; neoadjuvant therapy; chemotherapy; apatinib
MeSH Terms: conditions — Colonic Neoplasms | interventions — camrelizumab; apatinib; Drug Therapy

STUDY DESIGN:
Intervention Model Description: MSS/pMMR:Participants received 5 preoperative cycles of PD1 inhibitor and chemotherapy (mFOLFOX6), 2 months of apatinib, followed by surgery.
  Apatinib,PD1 inhibitor and chemotherapy needed to be stopped for 4-6 months before operation. 1 month after surgery, 7 cycles of mFOLFOX6 combined with PD-1 monoclonal antibody were performed as adjuvant therapy.
  MSI/dMMR:Participants received 5 preoperative cycles of PD1 inhibitor and 2 months of apatinib, followed by surgery.
  Apatinib,PD1 inhibitor needed to be stopped for 4-6 months before operation. 1 month after surgery, 7 cycles of PD-1 monoclonal antibody and apatinib were performed as adjuvant therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chemotherapy, PD-1 inhibitor and Apatinib (Experimental): Participants received 5 preoperative cycles of PD-1 inhibitor and chemotherapy (mFOLFOX6), 2 months of apatinib, followed by surgery. Apatinib,PD-1 inhibitor and chemotherapy needed to be stopped for 4-6 months before operation. 1 month after surgery, 7 cycles of mFOLFOX6 combined with PD-1 monoclonal antibody were performed as adjuvant therapy.
  Interventions: Drug: Camrelizumab , apatinib and chemotherapy

INTERVENTIONS:
Drug: Camrelizumab , apatinib and chemotherapy — Camrelizumab 200 mg, IV infusion on Days 1 each 14-day cycle
  Apatinib 250mg oral administration once a day, for two months
  mFOLFOX6 oxaliplatin 85 mg/m^2 IV infusion on Day 1 of each14-day cycle. Fluorouracil: 400 mg/m2 as a bolus injection given after a two-hour leucovorin infusion at a dose of 400 mg/m2. The loading dose is then followed by a 46-hour 5-fluorouracil infusion of 2,400 mg/m2 via a pump programmed to provide a constant drug infusion rate.

SUMMARY:
To determine the Efficacy and Safety of camrelizumab and apatinib combined with chemotherapy (mFOLFOX6) for MSS/pMMR locally advanced colon cancer.

DETAILED DESCRIPTION:
To determine the rate of tumor regression grade 2-4 at time of radical resection of MSS/pMMR colon cancer following neoadjuvant treatment.To determine the pathologic downstage rates at time of radical resection of colon cancer following neoadjuvant treatment, pathologic complete response (pCR) rates, R0 resection rate, 2 year Disease free survival, OS(overall survival) and adverse events, including perioperative complication and mortality rate.

To determine the pathologic downstage rates and pCR rate of radical resection of MSI/dMMR colon cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, ≤75 years
2. Histologically confirmed colon cancer ( tumor penetrated of muscularis propria depth ≥5mm of T3 , T4, N0-2, M0) without distant metastasis (AJCC 8th).
3. ECOG 0-1
4. Surgical treatment is planned after completion of neoadjuvant therapy
5. Patients can swallow pills normally
6. Expected overall survival ≥12 months
7. Blood routine: no blood transfusion or blood products usage within 14 days, G-CSF or other hematopoietic stimulator was not used. WBC counts > 3000/µl，Absolute neutrophil count (ANC) ≥ 1500 cells/µl，Platelet count ≥ 100,000/µl，Hemoglobin ≥ 9.0 g/dL.
8. AST, ALT and alkaline phosphatase ≤ 2.5 times the upper limit of normal (ULN)，Serum bilirubin ≤ 1.5 x ULN，creatinine<ULN
9. Prothrombin time (PT), international standard ratio (INR) ≤1.5 × ULN
10. Patients who have not received systemic chemotherapy or immunotherapy
11. Women of childbearing age must be willing to use adequate contraceptives during the study period of drug treatment;
12. Informed consent has been signed.

Exclusion Criteria:

1. Patients have received any prior systemic antitumor therapy;
2. Active bleeding within 3 months; Occurrence of arterial/venous thrombosis within 6 months; Hereditary or acquired bleeding (e.g., clotting dysfunction) or thrombotic tendencies; Full dose oral or injectable anticoagulants or thrombolytic drugs for therapeutic purposes are currently being used or have been used recently (10 days prior to the commencement of study treatment); Surgery (except for biopsy) was performed within 4 weeks prior to the study or the surgical incision was not fully healed; Aspirin (> 325 mg/ day) or dipyridamole, ticlopidine, clopidogrel, and silotazole are currently being used or have recently been used (10 days prior to the study).
3. Systemic corticosteroids or other systemic immunosuppressive drugs were used within 2 weeks prior to treatment. Immunosuppressive drugs were started or expected to be used during the trial. Inhaled corticosteroids, physiologic replacement doses of glucocorticoids are allowed.
4. Certain or suspected distant metastases.
5. The patient has a history of autoimmune disease.
6. Serious uncontrolled systemic diseases, such as severe active infections;
7. A person is known to be infected with the immunodeficiency virus (HIV) or known to be HIV-positive;
8. Patients have suffered from other malignancies in the past 5 years except cervical carcinoma in situ or basal cell carcinoma of the skin
9. Untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers (HBV DNA >500 IU/mL) or active HCV carriers with HCV RNA can be detected. Remarks: Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B patients (HBV DNA < 500 IU/mL) may be enrolled
10. Anti-infective therapy was not discontinued 14 days before the study;
11. A prior history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonia, and symptomatic interstitial lung disease or the presence of active pneumonia on a chest CT scan within 4 weeks prior to the study.
12. Patients have a history of intestinal obstruction within six months. Patients with incomplete obstruction syndrome of ileus at the time of initial diagnosis may be enrolled in the study if they have received definitive (surgical) treatment to resolve the symptoms, as assessed by the investigator.
13. Patients have non-resectable factors, including surgical contraindications
14. Patients Have high blood pressure that cannot be well controlled by antihypertensive medication (systolic ≥140 mmHg or diastolic ≥90 mmHg)
15. Urine routine indicated urinary protein ≥++ and confirmed 24-hour urinary protein >1.0g;
16. Known to be allergic to any study drug;
17. Patients have participated in other drug clinical studies within 4 weeks before enrollment;
18. Lactating women
19. According to the judgment of the researcher, the patient may have other factors that may affect the results of the study or cause the study to be terminated, such as alcohol abuse, drug abuse, other serious diseases (including mental diseases) requiring combined treatment. Patients have severe laboratory abnormalities, which will affect the safety of the patient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- First affiliated hospital, Zhejiang University, Hangzhou, Zhejiang, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy, PD-1 Inhibitor and Apatinib: Participants received 5 preoperative cycles of PD-1 inhibitor and chemotherapy (mFOLFOX6), 2 months of apatinib, followed by surgery. Apatinib,PD-1 inhibitor and chemotherapy needed to be stopped for 4-6 months before operation. 1 month after surgery, 7 cycles of mFOLFOX6 combined with PD-1 monoclonal antibody were performed as adjuvant therapy.
  Camrelizumab , apatinib and chemotherapy: Camrelizumab 200 mg, IV infusion on Days 1 each 14-day cycle
  Apatinib 250mg oral administration once a day, for two months
  mFOLFOX6 oxaliplatin 85 mg/m^2 IV infusion on Day 1 of each14-day cycle. Fluorouracil: 400 mg/m2 as a bolus injection given after a two-hour leucovorin infusion at a dose of 400 mg/m2. The loading dose is then followed by a 46-hour 5-fluorouracil infusion of 2,400 mg/m2 via a pump programmed to provide a constant drug infusion rate.
Period: Overall Study
Arm/Group | Chemotherapy, PD-1 Inhibitor and Apatinib
Started | 64
Completed | 12 (pCR 45.5% pMMR Patients, 87.5% patients had TRG 2-4)
Not Completed | 52

BASELINE CHARACTERISTICS:
Groups:
- Chemotherapy, PD-1 Inhibitor and Apatinib: From January 2021 to September 2022, 12 patients were enrolled. Most (10 [83.3%] of 12) patients were female. There were 10 patients (83.3%) with right-sided colon cancer. 7(58.3%) had cT4 stage tumors, and all patients had positive lymph nodes on baseline radiographic assessment. 10 (83.3%) completed the planned cycles of neoadjuvant therapy. 1 patient received 3 cycles of neoadjuvant therapy as a serious adverse event and 1 patient received 2 cycles of neoadjuvant therapy as tumor perforation . Of the 12 patients, 11 underwent surgery, of whom R0 resection was performed and 1 refused
Arm/Group | Chemotherapy, PD-1 Inhibitor and Apatinib
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
ECOG performance status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group performance status (ECOG PS) :The scale ranges from 0 to 5, with lower scores indicating better functioning.
  0. Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.
  Participants
    0 | 8
    1 | 3
    2 | 1
Clinical T stage [Count of Participants; unit: Participants] — T stage were staged using the 8th edition of the American Joint Committee of Cancer (AJCC) tumor-node-metastasis (TNM) staging classification for colon cancer.
  cT3:Tumor invades through the muscularis propria into pericolorectal tissues; cT4a:Tumor invades through the visceral peritoneum (including gross perforation of the bowel through tumor and continuous invasion of tumor through areas of inflammation to the surface of the visceral peritoneum); cT4b:Tumor directly invades or adheres to adjacent organs or structures
  Participants
    cT3 | 5
    cT4a | 5
    cT4b | 2
Clinical N stage [Count of Participants; unit: Participants] — cN0:No regional lymph node metastasis; cN1:One to three regional lymph nodes are positive (tumor in lymph nodes measuring ≥0.2 mm), or any number of tumor deposits are present and all identifiable lymph nodes are negative; cN2: Four or more regional lymph nodes are positive
  Participants
    cN0 | 0
    cN1 | 5
    cN2 | 7
MMR status [Count of Participants; unit: Participants] — pMMR:proficient mismatch repair; dMMR:deficiency in mismatch repair
  Participants
    dMMR | 4
    pMMR | 8

OUTCOME MEASURES:

1. Primary Outcome: Tumor Regression Rate of MSS/pMMR Patients
Description: the percentage of tumor regression rate (2-4) in pMMR patients
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Tumor Regression Grade Rate of pMMR Patients: the percentage of tumor regression rate (2-4) in pMMR patients
Arm/Group | Tumor Regression Grade Rate of pMMR Patients
Number analyzed (Participants) | 8
Participants | 7

2. Secondary Outcome: Pathologic Complete Response (pCR) Rates
Description: Percentage of patients with pathological complete response
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2025-12

3. Secondary Outcome: R0 Resection Rate
Description: R0 resection accounted for the percentage of all surgical patients=100%
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2025-12

4. Secondary Outcome: The Rate of 2 Year Disease Free Survival (DFS)
Description: Disease-free survival (DFS) is defined as the time from operation to recurrence of tumor or death. We will evaluate 2 year DFS is 100%
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2025-12

5. Secondary Outcome: Overall Survival (OS)
Description: Refers to the time of death from enrollment to any cause
Time Frame: 2 years
Reporting Status: Not Posted

6. Secondary Outcome: Event Free Survival (EFS)
Description: The period from the beginning of neoadjuvant therapy to the occurrence of any of the following events, whichever occurs first: tumor progression as assessed by RECIST 1.1; Tumor recurrence, including local recurrence or distant metastasis; Death from any cause; EFS=100%
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2025-12

7. Secondary Outcome: Perioperative Complication Rate
Description: The complication rate of all patients during the period around the time of a surgical operation
Time Frame: 3 months
Reporting Status: Not Posted

8. Secondary Outcome: Mortality Rate
Description: the ratio between deaths and all patients in the study during treatment
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Groups:
- Mortality Rate: the ratio between deaths and all patients in the study during treatment
Arm/Group | Mortality Rate
Number analyzed (Participants) | 12
Participants | 0

ADVERSE EVENTS:
Time Frame: 2 year
Description: Grade ≥3 adverse events occurred in 83.3% of patients, including neutropenia, decreased white blood cell count, thrombocytopenia, hypertension and alanine aminotransferase (ALT) increase.
Groups:
- Neutropenia: the most common adverse events were neutropenia (83.3%)
Arm/Group | Neutropenia
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 10/12
Other Adverse Events (participants affected / at risk) | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neutropenia (N=12)
neutropenia (Blood and lymphatic system disorders) | 10
decreased white blood cell count (Blood and lymphatic system disorders) | 4
thrombocytopenia (Blood and lymphatic system disorders) | 2
hypertension (Blood and lymphatic system disorders) | 2
ALT increased (Blood and lymphatic system disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neutropenia (N=12)
Hypertension (Cardiac disorders) | 2
RCCEP (Cardiac disorders) | 8
Vomiting (Gastrointestinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT04625803/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT04625803/SAP_001.pdf